CLINICAL TRIAL: NCT00359671
Title: Phase I Study Evaluating MK6592 in Combination With Docetaxel in Adult Patients With Relapsed or Refractory Advanced Solid Tumors
Brief Title: Treatment With MK6592 and an Anti-cancer Drug in Patients With Advanced Solid Tumors (6592-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6592-001; MK6592-001; 2006_508
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Advanced Solid Tumors

ARMS (2):
- 1 (Experimental): Arm 1: study drug
  Interventions: Drug: MK6592
- 2 (Other): Arm 2: study drug + comparator
  Interventions: Drug: MK6592; Drug: comparator: docetaxel

INTERVENTIONS:
Drug: MK6592 — MK6592 delivered as a 48-hour CIV as monotherapy in Cycle 1; 48-hour CIV of MK6592 in Cycle 2 and subsequent cycles.
Drug: comparator: docetaxel — docetaxel, delivered as a standard IV infusion.
  Arms: 2

SUMMARY:
A study to evaluate safety and tolerability of MK6592 in combination with an anti-cancer drug in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid tumors (metastatic or local) unresponsive to standard therapy, progressed on standard therapy, or no standard therapy exists. No limit to the number of prior treatment regimens
* Patients may be fully active without physical restrictions, ambulatory with restrictions on strenuous physical activity, or ambulatory and capable of self-care but not work activities (i.e., Eastern Cooperative Oncology Group performance status of greater than or equal to 2)
* Demonstrates adequate organ function (liver, kidneys, hematologic)

Exclusion Criteria:

* Chemotherapy or radiation therapy within 2 weeks of dosing; or unresolved side effects(s) from prior treatment regimen
* Participation in an investigational study within 14 days of dosing
* Primary central nervous system tumor
* Active brain or spinal cord metastases. Patients who completed a course of therapy for CNS metastases may be eligible if considered clinically stable for 3 months prior to study entry
* Symptoms from fluid in the abdomen or around the lungs
* Requires certain drugs or other products known to be metabolized by the liver enzyme CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MK6592 alone and in combination with docetaxel | 6 Months

SECONDARY OUTCOMES:
Observance of objective tumor responses in patients treated with MK6592 combined with docetaxel | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC